CLINICAL TRIAL: NCT00039039
Title: Phase III Randomized Study of Paclitaxel and Carboplatin or Cisplatin Followed by Radiotherapy With or Without Concurrent Paclitaxel in Patients With Unresectable Stage III Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy Followed by Radiation Therapy With or Without Paclitaxel in Treating Patients With Unresectable Stage III Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068846; INRC-PITCAP; EU-20202; INRC-ITA; NCI-V01-1665
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2006-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Drug Therapy; Cisplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: chemotherapy
Drug: cisplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as paclitaxel may make tumor cells more sensitive to radiation therapy. It is not yet known if combination chemotherapy followed by radiation therapy is more effective with or without paclitaxel in treating unresectable stage III non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy followed by radiation therapy with or without paclitaxel in treating patients who have unresectable stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival rate of patients with unresectable stage III non-small cell lung cancer treated with paclitaxel and carboplatin or cisplatin followed by radiotherapy with or without concurrent paclitaxel.
* Compare the 1-year survival rate and mean survival time in patients treated with these regimens.
* Compare the objective response rate and local control in patients treated with these regimens.
* Compare the tolerability of these regimens in these patients.
* Compare the safety profile and toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

All patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes or cisplatin IV on day 1. Treatment repeats every 21 days for 2 courses. Patients then proceed to randomized treatment.

* Arm I: Patients receive paclitaxel IV over 1 hour on day 1 and radiotherapy on days 1-5 of each week for 6 weeks.
* Arm II: Patients receive radiotherapy 5 days a week for 7 weeks. Patients are followed every 3 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 300 patients (150 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage III non-small cell lung cancer (NSCLC)

  * Locoregionally advanced unresectable disease
  * Previously untreated
* Measurable disease
* No involvement of supraclavicular lymph nodes
* No cytologically positive pleural or pericardial effusion
* No invasion to the wall of the esophagus or the cardiac ventricle
* No bone marrow involvement
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* WHO 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC greater than 4,000/mm^3
* Absolute neutrophil count greater than 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin less than upper limit of normal (ULN)
* AST and ALT less than 2.5 times ULN
* Alkaline phosphatase less than 5 times ULN
* No hepatic abnormalities

Renal:

* Creatinine less than ULN

Cardiovascular:

* No myocardial infarction within the past 6 months
* No cardiac insufficiency
* No uncontrolled arrhythmia

Pulmonary:

* FEV1 greater than 1 L
* DLCO at least 30% predicted
* No pneumonia
* No other non-disease-related pulmonary complications

Other:

* No more than 10% of total weight loss over the past 6 months
* No other disease that would preclude study
* No peripheral neuropathy grade 3 or greater
* No other prior or concurrent malignancy except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No familial, geographic, or psychological condition that would preclude study
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy
* No concurrent immunotherapy

Chemotherapy:

* No prior systemic chemotherapy

Endocrine therapy:

* No concurrent endocrine therapy

Radiotherapy:

* No prior radiotherapy for NSCLC

Surgery:

* See Disease Characteristics
* No prior complete resection of tumor
* Prior radical surgical resection allowed if local recurrence of disease
* No concurrent major surgery

Other:

* No other concurrent anticancer therapy or investigational agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2000-02

PRIMARY OUTCOMES:
Overall survival rate

SECONDARY OUTCOMES:
One-year survival rate and mean survival time
Objective response rate and local control
Tolerability
Safety profile, in terms of acute and delayed toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bruzzi, MD, MPH, PhD, Study Chair — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (37):
- Italy (37):
  - Ospedale Civile di Asti, Asti
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedali Riuniti di Bergamo, Bergamo
  - Spedali Civili di Brescia, Brescia
  - Civic Hospital of Carrara, Carrara
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Ospedale Mariano Santo, Cosenza
  - Azienda Istituti Ospitalieri, Cremona
  - Ospedale Santa Croce, Cuneo
  - Ospedale Galliera Oncologia, Genoa
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Ospedale San Martino, Genoa
  - Ospedale Civile di Ivrea, Ivrea
  - Ospedale Santa Maria Goretti, Latina
  - Ospedale Umberto I, Lugo DI Romagna
  - Istituto Policlinico San Donato, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milan
  - University of Modena Hospital and Reggio Emilia School of Medicine, Modena
  - Nuovo Ospedale San Gerardo at University of Milano-Bicocca, Monza
  - Azienda Ospedale S. Luigi at University of Torino, Orbassano
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Di Parma, Parma
  - Policlinico Monteluce, Perugia
  - Ospedale Santa Chiara Pisa, Pisa
  - Ospedale Sta. Maria Delle Croci, Ravenna
  - Ospedale Carlo Forlanini, Rome
  - Ospedale S. Camillo-Forlanini, Rome
  - Azienda Policlinico Umberto Primo, Rome
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
  - Istituto Regina Elena, Rome
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliera S. Maria, Terni
  - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Turin
  - Ospedale Evangelico Valdese, Turin
  - Ospedale Ostetrico Ginecologica Sant Anna, Turin
  - Azienda Ospedaliera Santa Maria della Misericordia, Udine
  - Ospedale San Bortolo, Vicenza